CLINICAL TRIAL: NCT04219917
Title: A Comparison of Kinesio® Taping Methods for Subjects With Patellar Tendonitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE20097
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Patellar Tendinitis
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hip (Experimental): Gluteus medius facilitation tape
  Interventions: Other: Kinesio Tape
- Knee (Experimental): Patellar sling tape
  Interventions: Other: Kinesio Tape
- Hip and Knee (Experimental): Gluteus medius facilitation and patellar sling tape
  Interventions: Other: Kinesio Tape

INTERVENTIONS:
Other: Kinesio Tape — Kinesio Tape will be applied to treat the pain associated with patellar tendonitis, to treat the cause of the pain, and to treat both factors.

SUMMARY:
The purpose of this study is to explore the possible effects Kinesio Tape may have on proprioception in individuals with patellar tendonitis. A supportive knee application, a facilitative hip application, and a combination of the two will be applied and compared. Within and between group comparisons will be drawn.

Participants will report for two research sessions with 24-36 hours between. Prior to arrival, they will complete a digital Victorian Institute of Sport Assessment for Patellar Tendonitis (VISA-P) and email it to the researcher. Participants must score less than 80 (out of a possible 100) to be considered for this study. If the individual meets the inclusion criteria, he/she will be scheduled for the 1st session. Upon arrival to the first session, informed consent will be obtained, the VISA-P will be reviewed, and intance of patellar tendonitis will be confirmed through palpation. Participants will then completed a Tampa Scale for Kinesiophobia (TSK) to measure fear of movement and a Visual Analog Scale (VAS) to measure overall pain. Height and weight measurments will be taken due to requirements of the Biodex Balance System (BBS), which will be used for balance measurements. Participants will take two, twenty-second practice tests, one with eyes open and one with eyes closed, followed by two minutes rest. Baseline testing will then be completed as follows: the participant will complete two tests with eyes open, and two tests with eyes closed on the injured leg, each with one minute rest between. The participant will then be taped with Kinesio Tape to either the hip, knee, or both the hip and knee according to the random group assignment. They will then rest for 15 minutes and complete a second round of balance testing with the same parameters as baseline testing. Participants will be scheduled for a second day no less that 24 hours and no more than 36 hours for re-test purposes.

On the second day of testing, participants will be given $10 for their participation on Day 1. If they want to continue with testing procedures, they will participate in the same balance testing procedures as Day 1. The integrety of the tape application will be confirmed, and second TSK and VAS scale will be administered. A final round of balance testing will be completed, and the participant will receive an additional $10 if they choose to complete both days of testing.

This research will allow us to compare results of the TSK, the VAS and the BBS testing both within subject and between group.

ELIGIBILITY:
Inclusion Criteria:

* score of less than 80 on the Victorian Institute of Sport Assessment for Patellar Tendonitis (VISA-P)
* experienced patellar tendon pain for greater than 14 days
* tender to palpation at the patellar tendon.

Exclusion Criteria:

* knee surgery in the last six months
* acute injury to the knee
* any pain in the ankles, hips or core that may compromise balance testing
* any allergy to adhesive
* malignancies
* cellulitis
* skin infection
* diabetes
* fragile skin

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Tampa Scale for Kinesiophobia | 24 hours
  Measures fear of movement, score range 17-68, higher score means higher degree of kinesiophobia
Visual Analog Scale | 24 hours
  Measures overall pain, score range 1-10, higher score indicates more pain
Biodex Balance System | 24 hours
  Measures balance

CONTACTS AND LOCATIONS:
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No